CLINICAL TRIAL: NCT03838588
Title: Tracking Genomic Cancer Evolution in Patients for Stage IB,II and IIIA Non-small Cell Lung Cancer After Radical Resection: The Tracking Molecular Evolution for NSCLC (T-MENC) Study
Brief Title: The Tracking Molecular Evolution for NSCLC (T-MENC) Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Geneplus-Beijing Co. Ltd. (Industry)
Collaborators: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Other Study IDs: T-MENC-NSCLC
Record Dates: First submitted 2019-02-10; First posted 2019-02-12 (Actual); Last update posted 2019-02-12 (Actual); Status verified 2019-02

CONDITIONS: Lung Neoplasms; Lung Cancer; Nonsmall Cell Lung Cancer; Adenocarcinoma of Lung
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Adenocarcinoma of Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood (including plasma, white cells), tissue.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- T-MENC Study Group: In the study, 200 of stage IB,II and IIIA non-small cell lung cancer patients obtained radical resection will be recruited. All the patients will receive biopsy genotype assay and ctDNA liquid biopsy. The abundance of mutations of ctDNA was tracked at 4 time points, including:
  1. st: 10 Days after patients received radical resection.
  2. nd: When patients finished the chemotherapy or target drug delivery two cycles.
  3. rd: 10 Days after patients finished the chemotherapy or target drug delivery four cycles.
  4. th: When tumor recrudescence / 2 years after radical resection. Tumor genomic clonal evolution was assessed by analyzing the relative abundance of mutations in plasma circulating tumor DNA (ctDNA).

SUMMARY:
Tumor genomic clonal evolution assessed with liquid biopsy of stage IB,II and IIIA non-small cell lung cancer patients after getting radical resection. Plasma circulating tumor DNA (ctDNA) analysis detects molecule residual disease and predicts recurrence in patients. The concordance of the relative abundance of mutations in plasma ctDNA with cancer recurrence.

DETAILED DESCRIPTION:
In the study, 200 of stage IB,II and IIIA non-small cell lung cancer patients obtained radical resection will be recruited. All the patients will receive biopsy genotype assay and ctDNA liquid biopsy. The abundance of mutations of ctDNA was tracked at 4 time points, including:

1. st: 10 Days after patients received radical resection.
2. nd: When patients finished the chemotherapy or target drug delivery two cycles.
3. rd: 10 Days after patients finished the chemotherapy or target drug delivery four cycles.
4. th: When tumor recrudescence / 2 years after radical resection.

Tumor genomic clonal evolution was assessed by analyzing the relative abundance of mutations in plasma circulating tumor DNA (ctDNA).

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent and assigned.
2. Newly diagnosed and histological or cytological confirmed stage IB-IIIA lung adenocarcinoma or non-smoking squamous cell carcinoma patients according to the AJCC staging system.
3. Expected radical resection.
4. Patients expected more than 3 months of survival time.
5. Willingness to comply with required protocols and give permission to use the data for clinical research and products development.

Exclusion Criteria:

1. Patients who want Neo-adjuvant therapy.
2. Patients with T3-4N1 Pancoast tumors (superior sulcal tumors).
3. Multi-station N2 non-small cell lung cancer with lymph node metastasis.
4. Eastern cooperative oncology group (ECOG) performance status > 2 after postoperative chemotherapy
5. Eastern cooperative oncology group (ECOG) performance status > 4 after postoperative targeted therapy.
6. Patients must never ever has received for any history of radiotherapy/ chemotherapy/surgery before.
7. Patients have other primary cancers.
8. Known central nervous system metastasis.
9. Patients expected less than 3 months of survival time.
10. Other situations mismatch this program.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Tracking Genomic Cancer Evolution in Patients for Stage IB,II and IIIA Non-small Cell Lung Cancer After Radical Resection.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-11-06 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Tumor genomic clonal evolution assessed with liquid biopsy of stage IB,II and IIIA non-small cell lung cancer patients after getting radical resection. | From assignment of the first subject to the time point when tumor recrudescence or 2 years after radical resection. The last participant will be recruited before June 30,2021.
  The tumor molecular clones and the frequency of gene mutations from 1021 tumor related genes will be detected by next-generation sequencing, which will be matched with the CT scanning.
The concordance of the plasma ctDNA detection status with Progress Free Survival (PFS) and Overall Survival (OS) after radical resection or/and under adjuvant therapy. | From assignment of the first subject to the time point when tumor recrudescence or 2 years after radical resection. The last participant will be recruited before June 30, 2021.
  Plasma circulating tumor DNA (ctDNA) analysis detects molecule residual disease and predicts recurrence in patients. All the patients will receive biopsy genotype assay and ctDNA liquid biopsy.

SECONDARY OUTCOMES:
Evaluation of ctDNA detecting assay in monitoring recurrence of early stage of lung cancer after radical resection. | From assignment of the first subject to the time point when tumor recrudescence or 2 years after radical resection. The last participant will be recruited before June 30, 2021.
  All the patients will receive biopsy genotype assay and ctDNA liquid biopsy.
The molecular mechanism between the tumor recurrence and ctDNA mutations | From assignment of the first subject to the time point when tumor recrudescence or 2 years after radical resection. The last participant will be recruited before June 30, 2021.

CONTACTS AND LOCATIONS:
Overall Officials: Yi Zhang, MD, Study Chair — Xuanwu Hospital, Beijing; Yao guang Sun, MD, Principal Investigator — Beijing Hospital; Jie Li, MD, Principal Investigator — Beijing Friendship Hospital, Capital Medical University, Beijing 100050, China +86-139 1189 2587 lijie821cn@163.com; Hong Zhang, MD, Principal Investigator — The First Hospital of Jilin University; Zhi qiang Wang, MD, Principal Investigator — Tangshan People's Hospital; Ming He, MD, Principal Investigator — Beijing Chest Hospital, Capital Medical University; Zi dan Wang, MD, Principal Investigator — Beijing Chest Hospital, Capital Medical University; Li jun Liu, MD, Principal Investigator — Hebei General Hospital; Kang Shao, MD, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences; Chao yang Liang, Principal Investigator — China-Japan Friendship Hospital
Locations (10):
- China (10):
  - Beijing Hospital, Beijing, Beijing Municipality
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - China-Japan Friendship Hospital, Beijing, Beijing Municipality
  - Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Xuanwu Hospital Capital Medical University, Beijing, Beijing Municipality
  - Beijing Chest Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Hebei General Hospital, Shijiazhuang, Hebei
  - Tangshan People's Hospital, Tangshan, Hebei
  - The First Bethune Hospital of Jilin University, Changchun, Jilin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bettegowda C, Sausen M, Leary RJ, Kinde I, Wang Y, Agrawal N, Bartlett BR, Wang H, Luber B, Alani RM, Antonarakis ES, Azad NS, Bardelli A, Brem H, Cameron JL, Lee CC, Fecher LA, Gallia GL, Gibbs P, Le D, Giuntoli RL, Goggins M, Hogarty MD, Holdhoff M, Hong SM, Jiao Y, Juhl HH, Kim JJ, Siravegna G, Laheru DA, Lauricella C, Lim M, Lipson EJ, Marie SK, Netto GJ, Oliner KS, Olivi A, Olsson L, Riggins GJ, Sartore-Bianchi A, Schmidt K, Shih lM, Oba-Shinjo SM, Siena S, Theodorescu D, Tie J, Harkins TT, Veronese S, Wang TL, Weingart JD, Wolfgang CL, Wood LD, Xing D, Hruban RH, Wu J, Allen PJ, Schmidt CM, Choti MA, Velculescu VE, Kinzler KW, Vogelstein B, Papadopoulos N, Diaz LA Jr. Detection of circulating tumor DNA in early- and late-stage human malignancies. Sci Transl Med. 2014 Feb 19;6(224):224ra24. doi: 10.1126/scitranslmed.3007094. PMID 24553385
- [Result] Tie J, Wang Y, Tomasetti C, Li L, Springer S, Kinde I, Silliman N, Tacey M, Wong HL, Christie M, Kosmider S, Skinner I, Wong R, Steel M, Tran B, Desai J, Jones I, Haydon A, Hayes T, Price TJ, Strausberg RL, Diaz LA Jr, Papadopoulos N, Kinzler KW, Vogelstein B, Gibbs P. Circulating tumor DNA analysis detects minimal residual disease and predicts recurrence in patients with stage II colon cancer. Sci Transl Med. 2016 Jul 6;8(346):346ra92. doi: 10.1126/scitranslmed.aaf6219. PMID 27384348
- [Result] Abbosh C, Birkbak NJ, Wilson GA, Jamal-Hanjani M, Constantin T, Salari R, Le Quesne J, Moore DA, Veeriah S, Rosenthal R, Marafioti T, Kirkizlar E, Watkins TBK, McGranahan N, Ward S, Martinson L, Riley J, Fraioli F, Al Bakir M, Gronroos E, Zambrana F, Endozo R, Bi WL, Fennessy FM, Sponer N, Johnson D, Laycock J, Shafi S, Czyzewska-Khan J, Rowan A, Chambers T, Matthews N, Turajlic S, Hiley C, Lee SM, Forster MD, Ahmad T, Falzon M, Borg E, Lawrence D, Hayward M, Kolvekar S, Panagiotopoulos N, Janes SM, Thakrar R, Ahmed A, Blackhall F, Summers Y, Hafez D, Naik A, Ganguly A, Kareht S, Shah R, Joseph L, Marie Quinn A, Crosbie PA, Naidu B, Middleton G, Langman G, Trotter S, Nicolson M, Remmen H, Kerr K, Chetty M, Gomersall L, Fennell DA, Nakas A, Rathinam S, Anand G, Khan S, Russell P, Ezhil V, Ismail B, Irvin-Sellers M, Prakash V, Lester JF, Kornaszewska M, Attanoos R, Adams H, Davies H, Oukrif D, Akarca AU, Hartley JA, Lowe HL, Lock S, Iles N, Bell H, Ngai Y, Elgar G, Szallasi Z, Schwarz RF, Herrero J, Stewart A, Quezada SA, Peggs KS, Van Loo P, Dive C, Lin CJ, Rabinowitz M, Aerts HJWL, Hackshaw A, Shaw JA, Zimmermann BG; TRACERx consortium; PEACE consortium; Swanton C. Phylogenetic ctDNA analysis depicts early-stage lung cancer evolution. Nature. 2017 Apr 26;545(7655):446-451. doi: 10.1038/nature22364. PMID 28445469
- [Result] Chaudhuri AA, Chabon JJ, Lovejoy AF, Newman AM, Stehr H, Azad TD, Khodadoust MS, Esfahani MS, Liu CL, Zhou L, Scherer F, Kurtz DM, Say C, Carter JN, Merriott DJ, Dudley JC, Binkley MS, Modlin L, Padda SK, Gensheimer MF, West RB, Shrager JB, Neal JW, Wakelee HA, Loo BW Jr, Alizadeh AA, Diehn M. Early Detection of Molecular Residual Disease in Localized Lung Cancer by Circulating Tumor DNA Profiling. Cancer Discov. 2017 Dec;7(12):1394-1403. doi: 10.1158/2159-8290.CD-17-0716. Epub 2017 Sep 24. PMID 28899864